CLINICAL TRIAL: NCT06956742
Title: Effect of Intermittent Intrapulmonary Deflation on the Sensory Dimension of Dyspnea After Exercise in Patients With Chronic Obstructive Pulmonary Disease: A Double-blind, Randomized Crossover Study
Brief Title: Intermittent Intrapulmonary Deflation and Dyspnea Following Exercise in People With Chronic Obstructive Pulmonary Disease
Acronym: DEFLA-DYSPNEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Collaborators: PhysioAssist (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: DEFLA-DYSPNEA
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic obstructive pulmonary disease; Intermittent intrapulmonary deflation; Dypsnea; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single-center, randomized controlled, prospective, two-arm crossover trial with concealed allocation and double-blinding (participants and evaluators).
  This study will be accompanied by a pre-planned ancillary study designed to evaluate the acute effects of using the intermittent intrapulmonary deflation device on the same outcomes, based on the initial randomization sequence at the first visit (see Study Description section). Consequently, this ancillary study is a single-center, randomized controlled, prospective, parallel trial with concealed allocation and double blinding (participants and evaluators).
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active intermittent intrapulmonary deflation (Experimental): One week home-based treatment period.
  Interventions: Device: Active intermittent intrapulmonary deflation.
- Placebo intermittent intrapulmonary deflation (Placebo Comparator): One week home-based treatment period.
  Interventions: Device: Placebo intermittent intrapulmonary deflation.

INTERVENTIONS:
Device: Active intermittent intrapulmonary deflation. — Intermittent intrapulmonary deflation sessions will be performed using the SIMEOX device (SIMEOX, PhysioAssist, Aix-en-Provence, France), which will be delivered to the patient's home by a home healthcare provider. The device power setting (25%, 50%, 75%, or 100%) will be individualized according to the parameters determined during the familiarization visit by a trained physiotherapist. Patients will be instructed to perform tidal volume inspirations followed by passive expirations into the device through a mouthpiece, up to their maximal tolerance. The device will be activated by the patient during expiration using a manual remote control.
  Each device usage cycle consists of 10 expirations, with oscillations generated at 12 Hz during the first 8 cycles and at 6 Hz during the last 2 cycles. Rest periods will be allowed during the session, and a mandatory pause will be imposed every 10 expirations. The session duration is fixed at 20 minutes, with patients performing one session in the
  Arms: Active intermittent intrapulmonary deflation
Device: Placebo intermittent intrapulmonary deflation. — Placebo intermittent intrapulmonary deflation sessions will be performed using the SIMEOX device (SIMEOX, PhysioAssist, Aix-en-Provence, France), which will be delivered to the patient's home by a home healthcare provider. Due to the physiological mechanism of action of the device (intermittent negative pressure with increasing intensity, inversely proportional to airflow resistance), it is assumed that device use under placebo conditions will be infra-therapeutic.
  To ensure this, the device will be set to the same setting as the active intermittent intrapulmonary deflation session but an intentional air leak will be introduced into the circuit at the device's output (not visible to the participant) to prevent the generated negative pressure from exceeding t The validity of this placebo condition will be confirmed through bench tests.
  All other conditions will remain identical to the active intermittent intrapulmonary deflation sessions. Patients will be instructed to perform tidal vo
  Arms: Placebo intermittent intrapulmonary deflation

SUMMARY:
Chronic obstructive pulmonary disease is a long-term lung condition that causes breathing difficulties. People living with this disease often feel short of breath, especially during physical activity, which can make daily tasks more challenging. This breathlessness is partly caused by mucus accumulation within the airways and air getting trapped in the lungs. Both of these reduce the amount of fresh air that can enter with each breath and increase the effort required to breathe.

To manage symptoms, people with chronic obstructive pulmonary disease may use medications, oxygen therapy, or be referred to pulmonary rehabilitation programs. These programs often include exercise training, self-management strategies, and airway clearance techniques. While chest physiotherapists typically guide patients in these techniques, certain medical devices can also help individuals manage their condition independently at home.

One such device uses a method called intermittent intrapulmonary deflation, which involves applying gentle pressure changes through a mouthpiece to help loosen mucus and release trapped air from the lungs. Although some individuals already use this kind of device as part of their daily care, more scientific evidence is needed to determine whether the improvements in airway clearance and reduced air trapping actually lead to measurable relief of breathlessness.

The goal of this clinical trial is to find out whether this type of medical device designed to remove airway mucus and trapped air in the lungs (using intermittent intrapulmonary deflation) can help reduce breathlessness (dyspnea) after physical activity in people with COPD.

The main questions this study aims to answer are:

* Does using the device at home for one week reduce the intensity of breathlessness after walking?
* Does it also improve walking distance, reduce the feeling of muscle fatigue, or increase satisfaction with the airway clearance method?

Researchers will compare the active device to a placebo device that looks and feels identical but does not deliver the active treatment. This comparison will help determine whether the observed effects are due to the device itself or other factors such as expectations or chance.

Participants in this study will be adults diagnosed with moderate to very severe chronic obstructive pulmonary disease. All participants must have recently completed a pulmonary rehabilitation program, continue to experience breathlessness while walking, and show signs of lung hyperinflation (when air remains trapped in the lungs). People will not be included if they have other serious health conditions that could make walking difficult or unsafe, or if they have any contraindications to using the device.

Participants who agree to participante in the study will:

* Attend a visit at the pulmonary rehabilitation center for baseline testing and to learn how to use the device;
* Be randomly assigned to use either the active device or the placebo device at home for 7 days;
* Return to the center for walking tests, lung function tests, and questionnaires about breathing and fatigue;
* After a one-week break, use the device with alternative settings (the one not used in the first phase) for another 7 days;
* Complete a final visit at the end of the study to repeat the same tests.

Participants will also be invited to take part in an ancillary study during their first clinic visit to examine how a single session with the device affects breathlessness immediately after walking.

This research will help determine whether this non-pharmacological, device-based method of clearing mucus and reducing trapped air can bring meaningful improvement in breathlessness for people with chronic obstructive pulmonary disease, especially when used at home. If effective, it may offer a simple and convenient way to help people breathe more comfortably during everyday activities.

Participants will receive compensation for their time and travel.

DETAILED DESCRIPTION:
Dyspnea in chronic obstructive pulmonary disease is multifactorial and results from complex pathophysiological mechanisms. A key contributor is dynamic hyperinflation, caused by airflow obstruction and expiratory airway collapse during exertion. Excessive mucus production and impaired mucociliary clearance further contribute to airway obstruction, yet mucus management remains an underexplored therapeutic target.

Current airway clearance techniques, such as manual chest physiotherapy and positive expiratory pressure devices, often require forced expiration and primarily act on proximal airways. In contrast, intermittent intrapulmonary deflation is a novel approach applying intermittent negative pressure during expiration to facilitate secretion mobilization, potentially improving expiratory flow and reducing lung hyperinflation. Intermittent intrapulmonary deflation is active only during passive exhalation, can be self-administered at home, and may provide an alternative for patients chronic pulmonary disease who experience chronic mucus retention.

This study aims to assess the effect of intermittent intrapulmonary deflation on dyspnea after exercise in individuals with chronic obstructive pulmonary disease. By improving secretion clearance and reducing dynamic hyperinflation, intermittent intrapulmonary deflation could represent a novel strategy to alleviate dyspnea, enhance exercise tolerance, quality of life, and address a significant unmet clinical need in this population.

Primary objective: to evaluate the effect of using an intermittent intrapulmonary deflation device for one week at home on the sensory dimension of dyspnea after exercise in individuals with chronic obstructive pulmonary disease.

Secondary objectives: to evaluate the effect of using an intermittent intrapulmonary deflation device for one week at home on exercise capacity, dyspnea perception (affective dimension and dyspnea intensity), perception of lower limb muscle fatigue, breathing pattern, operational lung volume, critical inspiratory constraints, and heart rate measured at the end of exercise. Additionally, the study aims to assess the depth of oxygen desaturation during exercise, participant satisfaction, respiratory function, and adverse events.

This is a prospective, randomized, controlled, double-blind, crossover clinical trial conducted in a single center, with concealed allocation. Participants will undergo two 7-day intervention periods at home (active or placebo device), separated by a minimum of 7days (maximum 28 days) washout phase. Each participant will serve as their own control.

This study will be accompanied by a pre-planned ancillary study designed to evaluate the acute effects of using the intermittent intrapulmonary deflation device on the same outcomes, based on the initial randomization sequence at the first visit. Consequently, this ancillary study is a single-center, randomized controlled, prospective, parallel trial with concealed allocation and double blinding (participants and evaluators).

This clinical trial comprises six phases: an initial visit (visit 1) at the pulmonary rehabilitation center, a one-week home-based treatment period utilizing either the investigational device or the placebo device, an intermediate visit after this first week (visit 2), a washout period (minimum one week, maximum 4 four weeks), a subsequent one-week home-based treatment period with the alternative condition, and a final visit at the center (visit 3). Further details about de content of these visit are available below.

Inclusion visit (visit 1):

The visit is conducted by the recruitment officer who also verifies the patient's eligibility criteria. The recruitment officer also informs the patient and answers all questions regarding the objective, nature of constraints, foreseeable risks, and expected benefits of the clinical investigation. They specify the patient's rights in the context of the clinical investigation and provide a copy of the information note and consent form to the patient.

Before any examination related to the clinical investigation, the recruitment officer obtains the patient's free, informed, and written consent.

This visit follows the 14 steps described below. Steps 8 to 14 belong to a pre-planned ancillary clinical investigation aimed at examining the acute effects of using an intermittent intrapulmonary deflation device on the sensory dimension of dyspnea and other outcomes after exertion, in individuals with chronic obstructive pulmonary disease.

1. Information, written consent, and collection of demographic data;
2. Assessment of dyspnea at rest, health status, and quality of life;
3. Evaluation of respiratory function and breathing pattern at rest in a seated position;
4. Installation of a pulse oximeter and performance of a six-minute walk test, with the patient's usual oxygen flow rate;
5. Post-exercise assessment: dyspnea and muscle fatigue of the lower limbs, breathing pattern, operational lung volume, and critical inspiratory constraints;
6. Familiarization and training on the use of the intermittent intrapulmonary deflation device (SIMEOX, PhysioAssist, Aix-en-Provence, France), and determination of the optimal setting by the operator (device power percentage ranging from 25 to 100% to reach the clinical efficacy indicator); the operator informs the patient that different settings are being studied during the clinical investigation without further details and does not provide indications regarding the clinical efficacy indicator; the operator also ensures that the patient is capable of performing deep and maximal inspiratory maneuvers. This initiation should be time-limited to avoid representing a complete session to minimize any physiological effects.
7. Randomisation.

   Pre-planned ancilliary clinical investigation:
8. Assessment of dyspnea ;
9. Performance a single 20-minute session with the intermittent intrapulmonary deflation device or with the placebo, according to the randomisation sequence;
10. Assessment of dyspnea and muscle fatigue of the lower limbs;
11. Evaluation of respiratory function and breathing pattern;
12. Installation of a pulse oximeter and performance of the six-minute walk test by an evaluator unaware of the allocation, with the patient's usual oxygen flow rate;
13. Post-exercise assessment: dyspnea and muscle fatigue of the lower limbs, breathing pattern, operational volume, and critical inspiratory constraints;
14. Assessment of participant's satisfaction.

At the end of this visit, a home healthcare provider will provide the intermittent intrapulmonary deflation device for one week. Patients are invited to use the device independently at home according to the randomization sequence, for 20 minutes, twice daily. A phone appointment is scheduled for the first day of independent use and on the fourth day. Any identified difficulties in use will lead to the scheduling of another appointment the following day.

Follow-up visit at the end of the first sequence (visit 2):

The visit is conducted by the evaluator, who is unaware of the patient's allocation. The details of this visit are described below:

1. Assessment of dyspnea and muscle fatigue of the lower limbs;
2. Evaluation of respiratory function and breathing pattern, at rest in a seated position;
3. Installation of a pulse oximeter and performance of the six-minute walk test by an evaluator unaware of the order in which the patient used the device, with the patient's usual oxygen flow rate;
4. Post-exercise assessment: dyspnea and muscle fatigue of the lower limbs, breathing pattern, operational volume, and critical inspiratory constraints;
5. Assessment of participant satisfaction.

Washout period:

After the second visit, patients are asked not to use the device for at least one week (maximum four weeks). This is ensured by providing a limited number of consumables that will not allow device use beyond the first week.

At the end of this washout period, the home healthcare provider will return to the patient's home to equip them with the device required for the alternative condition, according to the randomization sequence.

Follow-up visit at the end of the second sequence (visit 3) and conclusion of the research:

The visit is conducted by the evaluator, who is unaware of the patient's allocation. This visit strictly follows the same procedures as visit 2.

At the end of this visit, the research is considered completed, and the home healthcare provider retrieves the device provided to the patient's home.

Randomisation and interventions: the sequence for administering the therapeutic modalities (active device followed by placebo, or placebo followed by active device) will be determined randomly using a computer-generated list (randomizer.org) in alternating blocks of 4 and 6, with a 1:1 ratio. The block sizes will remain undisclosed to the recruiting operator to prevent bias. This list will be maintained by an individual external to the study, who will be contacted by the recruitment operator during patient inclusion to determine the allocation sequence (concealed allocation). A document detailing the randomisation procedure will be kept confidential at the sponsor site.

* Sequence A: active device → washout → placebo device
* Sequence B: placebo device → washout → active device

Active intermittent intrapulmonary deflation sessions will be performed using the SIMEOX device (SIMEOX, PhysioAssist, Aix-en-Provence, France), which will be delivered to the patient's home by a home healthcare provider. The device power setting (25%, 50%, 75%, or 100%) will be individualized according to the parameters determined during the familiarization visit (visit 1). Patients will be instructed to perform tidal volume inspirations followed by passive expirations into the device through a mouthpiece, up to their maximal tolerance. The device will be activated by the patient during expiration using a manual remote control.

Each device usage cycle consists of 10 expirations, with oscillations generated at 12 Hz during the first 8 cycles and at 6 Hz during the last 2 cycles. Rest periods will be allowed during the session, and a mandatory pause will be imposed every 10 expirations. The session duration is fixed at 20 minutes, with patients performing one session in the morning and another in the afternoon or evening.

Placebo intermittent intrapulmonary deflation sessions will be performed using the SIMEOX device (SIMEOX, PhysioAssist, Aix-en-Provence, France), which will be delivered to the patient's home by a home healthcare provider. Due to the physiological mechanism of action of the device (intermittent negative pressure with increasing intensity, inversely proportional to airflow resistance), it is assumed that device use under placebo conditions will be infra-therapeutic.

To ensure this, the device will be set to the same power setting as the active intermittent intrapulmonary deflation session but an intentional air leak will be introduced into the circuit at the device's output (not visible to the participant) to prevent the generated negative pressure from exceeding the minimum effective threshold. The validity of this placebo condition will be confirmed through bench tests.

All other conditions will remain identical to the active intermittent intrapulmonary deflation sessions. Patients will be instructed to perform tidal volume inspirations, followed by passive expirations into the device through a mouthpiece, up to their maximal tolerance. The device will be activated by the patient during expiration using a manual remote control.

Each device usage cycle will consist of 10 expirations, with oscillations generated at 12 Hz during the first 8 cycles and at 6 Hz during the last 2 cycles. Rest periods will be allowed during the session, with a mandatory pause every 10 expirations. The session duration is fixed at 20 minutes, with patients performing one session in the morning and another in the afternoon or evening.

Blinding of the evaluator: evaluations will be conducted by an assessor who is blinded to the order in which the patient has used the device. Data will be recorded in an electronic data collection form (Dotter.Science, KerNel Biomedical) by the assessor, who will remain unaware of the intervention.

Blinding of the participant: due to the physiological mechanism of the device (intermittent negative pressure increasing with resistance to airflow), it is assumed that the use of the device in the placebo condition will be sub-therapeutic. To achieve this, the device will be set to a low power for all participants, and a deliberate leak will be incorporated into the output circuit (invisible to the participant) to ensure that the maximum pressure achieved is below the effective minimum negative pressure (-10 cm H2O). The validity of this placebo condition will be confirmed in advance through bench tests. The remaining modalities will mirror those of the active intermittent intrapulmonary deflation session.

Blinding of the statistician: statistical analyses plan will be defined a priori. Statistical analysis will be conducted by an independent statistician who will be unaware of the randomization sequence.

Sample size calculation for a superiority study based on the primary outcome (sensory dimension of dyspnea assessed using the multidimensional dyspea profile questionnaire): to detect a mean difference of at least 2 points between interventions (corresponding to the established minimal clinically important difference for the primary outcome), and considering a moderate effect size of 0.5, a type I error rate of 5%, and a power of 80%, a total of 33 participants will be required. Accounting for a 15% loss to follow-up, up to 40 participants may be included (20 in each crossover group) to ensure that 33 participants have an available measurement for the primary outcome.

Statistical analysis :

Analysis populations:

Three analysis populations will be involved in this study:

* The full analysis Sst will include all randomized participants with at least one efficacy assessment. For those who do not complete the treatment as planned, the last observation will be used as the final outcome (last observation carried forward).
* The per protocol set will include all randomized participants who completed all visits in accordance with the protocol.
* The adherent population will include all randomized participants who completed at least 70% of the prescribed sessions, which is defined 10 sessions or more.

Description of the population:

Qualitative variables will be described by counts and frequencies. Quantitative variables will be summarized using means, standard deviations, and when justified by the distribution of the variable, medians and quartiles will also be reported.

Analysis of outcomes measured only at the end of exercise (performance during the six-minute walk test, nadir transcutaneous oxygen saturation, etc.):

A mixed linear model will be employed for each outcome. The values obtained during the first 6MWT (at rest before the test when available, and after the test), the order of the tests (first or second test), the sequence order (active first then placebo, or placebo first then active), and the treatment modality (active or placebo) will be included as fixed effects, with the participant included as a random effect.

Analysis of other outcomes:

A mixed linear model will be utilized for each outcome. The values obtained during the first six-minute walk test at rest before the test when available, and after the test, and after exercise), the order of the tests (first or second test), the sequence order (active first then placebo, or placebo first then active), the treatment modality (active or placebo), the time of measurement (baseline or post-exercise), and the interaction between treatment modality and time of measurement will be included as fixed effects, with the participant as a random effect.

Analysis of ancillary study endpoints:

The ancillary study will also focus on the primary endpoint and secondary endpoints measured before and/or after the 6MWT, after randomization. A mixed linear model or a mixed logistic model will be used. In this model, the treatment modality (active or placebo) and values obtained during the first 6MWT at inclusion will be included as fixed effects, with the participant as a random effect for variables collected only at the end of exercise. For values measured before and after exercise, the time of measurement (baseline or post-exercise) and the interaction between treatment modality and time of measurement will also be included as fixed effects.

Note 1: the values obtained during the first 6MWT at inclusion are the values at inclusion for each criterion before and after the 6MWT at inclusion. For example, for the primary endpoint, we will use the values of the sensory dimension of dyspnea at inclusion (at rest before the test, and at the end of the test).

Note 2: Statistical models may take into account the interaction between treatment modality and treatment sequence.

The effect of intermittent intrapulmonary pressure release on the proportion of patients with a desaturation of ≥4% will be studied using the McNemar test.

Presentation of results Data will be reported as mean differences (95% confidence intervals) and interpreted according to the minimal clinically important difference for each criterion (when available in the literature) or based on the clinical expertise of the investigators.

Secondary analysis A dose-response analysis will be conducted. The number of sessions will be considered as the dose and the primary endpoint as the response.

Sensitivity analysis A sensitivity analysis will be conducted to assess the influence of various factors, such as the use of inhaled treatments (all types of bronchodilators and anticholinergics), GOLD stage, the presence or absence of oxygen therapy and/or non-invasive ventilation, participant age, or secretory phenotype (based on a COPD Assessment Test score ≥ 6 from the sum of questions 1 and 2, or the Saint George's Respiratory Questionnaire score).

Analyses will be performed using GraphPad Prism 8 and R software.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* COPD stage GOLD II to IV;
* Completion of a pulmonary rehabilitation program within the last 6 months;
* 6-minute walk test < 350 meters before and/or after completing the pulmonary; rehabilitation program;
* mMRC dyspnea scale ≥ 2;
* Pulmonary hyperinflation (ratio between residual volume to total lung capacity superior to 50%, and either total lung capacity superior to 130% or functional residual capacity superior to 130%);
* With or without oxygen supplementation;
* Stable condition (no exacerbation or change in treatment in the last 4 weeks);
* Naïve to intermittent intrapulmonary deflation.
* Regulatory criteria (social security affiliation; adult patient who has read and understood the information letter and signed the informed consent form).

Non-inclusion Criteria:

* Pregnant women or likely to be;
* Patients under guardianship or curatorship;
* Inability to consent;
* Primary diagnosis of another chronic obstructive respiratory disease such as asthma or primary bronchiectasis;
* Orthopedic, neurological, vascular, or neuromuscular conditions that limit walking or require walking aids;
* Severe or unstable cardiovascular disease (uncontrolled cardiac arrhythmias, severe heart failure, recent myocardial infarction, unstable angina);
* Patients actively requiring assistance with inspiration (e.g. ventilatory assistance with endotracheal tube, tracheostomy tube, or ventilated with a mask; patients with neuromuscular disease with respiratory muscle weakness; patients with inability to cough forcefully and independently);
* Hemodynamic instability;
* Recent pneumothorax (within the last 3 months);
* Recent pulmonary or upper airway surgery (within the last month);
* Referral to a pulmonary rehabilitation program in preparation for thoracic surgery (lung volume reduction, lung transplantation, or lung resection for non-small cell lung cancer);
* Use of an electrical mechanical device for airway clearance during the study period (in-exsufflator, high-frequency chest oscillation, etc.);
* Active cancer;
* Severe episode of hemoptysis in the last 3 months;
* Severe tracheomalacia.

Exclusion Criteria:

* Withdrawal of consent;
* Acute COPD exacerbation between visits or onset of cardiorespiratory instability;
* Use of an electrical mechanical device for airway clearance during the study period (in-exsufflator, high-frequency chest oscillation, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Sensory dimension of dyspnea | Day 8 (after seven days of intervention)
  The sensory dimension of dyspnea will be assessed using French version of the Multidimensional Dyspnea Profile questionnaire, taking into account the last 30 seconds of effort during the 6-minute walk test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a greater sensory dimension of dyspnea. The established minimal clinically important difference for this outcome is 2 points.

SECONDARY OUTCOMES:
Functional exercise capacity - Six-minute walk test | Day 8 (after seven days of intervention).
  Functional exercise capacity will be evaluated using the 6-minute walk test. It will be conducted following the guidelines of the American Thoracic Society and the European Respiratory Society. Patients will be instructed to cover the maximum distance possible within 6 minutes. The test will be performed in a corridor with a minimum length of 30 meters. The established minimal clinically important difference for this test is 25 meters.
Affective dimension of dyspnea | Day 8 (after seven days of intervention).
  The affective dimension of dyspnea will be assessed using the french version of the Multidimensional Dyspnea Profile questionnaire, considering the last 30 seconds of effort during the 6-minute walk test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a significant affective dimension of dyspnea. The established minimal clinically important difference for this outcome is 3 points.
Intensity of dyspnea | Day 8 (after seven days of intervention).
  The intensity of dyspnea will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of your breathlessness?" The minimal clinically important difference for this outcome is 1 point. Outcome will be assessed at the end of the six-minute walk test.
Intensity of lower limb fatigue | Day 8 (after seven days of intervention).
  The intensity of muscle fatigue in the lower limbs will be assessed using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of fatigue) and 10 (maximal fatigue). Patients will be asked, "What is the intensity of the fatigue in your legs?" The minimal clinically important difference for this outcome is 1 point. Outcome will be assessed at the end of the six-minute walk test.
Respiratory function - Forced expiratory volume in 1 second | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Vital capacity | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Forced vital capacity | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Ratio between forced expiratory volume in 1 second to forced vital capacity | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France).
Respiratory function - Functional residual capacity | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Total lung capacity | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Residual volume | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Airway resistance | Day 8 (after seven days of intervention).
  Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France).
Breathing pattern - Tidal volume | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Respiratory rate | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Inspiratory time | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Expiratory time | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Ratio between inspiratory time to expiratory time | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Minute ventilation | Day 8 (after seven days of intervention).
  Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds. Minute ventilation will be calculated as the product of tidal volume and respiratory rate.
Operational lung volume - Inspiratory capacity | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Operational lung volume - End inspiratory lung volume | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  End inspiratory lung volume will be calculated as total lung capacity - inspiratory capacity + tidal volume.
Operational lung volume - End expiratory lung volume | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  End expiratory lung volume will be calculated as total lung capacity - inspiratory capacity.
Critical inspiratory constraints - Ratio between tidal volume to inspiratory capacity | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Critical inspiratory constraints - Ratio between tidal volume to vital capacity | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Critical inspiratory constraints - Inspiratory reserve volume | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  Inspiratory reserve volume will be calculated as inspiratory capacity - tidal volume.
Critical inspiratory constraints - Ratio between inspiratory reserve volume to total lung capacity | Day 8 (after seven days of intervention).
  Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Transcutaneous oxygen saturation during a six-minute walk test | Day 8 (after seven days of intervention).
  Transcutaneous oxygen saturation (SpO₂) will be measured at rest and continuously throughout the 6-minute walk test using a pulse oximeter (Nonin WristOx2 3150, Nonin Medical Inc., Plymouth, MN, USA). Data collection will be performed using Nvision software (Henrotch, Aartselaar, Belgium). The SpO₂ value at the end of the test, as well as the nadir SpO₂ (lowest recorded value) during the 6MWT, will be reported. The proportion of patients experiencing oxygen desaturation ≥ 4%, as well as the proportion of patients with desaturation ≥ 4% and SpO₂ < 90%, will also be documented. Finally, the total time spent with SpO₂ < 90% will be analyzed.
Heart rate during the six-minute walk test | Day 8 (after seven days of intervention).
  Heart rate will be measured at rest and continuously throughout the six minute xalk test using a pulse oximeter (Nonin WristOx2 3150, Nonin Medical Inc., Plymouth, MN, USA). Data collection will be performed using Nvision software (Henrotch, Aartselaar, Belgium). The highest HR recorded during the test and the HR at the end of the test will be reported.
Patient satisfaction | Day 8 (after seven days of intervention).
  Patient satisfaction will be assessed using a visual analog scale ranging from 0 (not satisfied at all) to 10 (extremely satisfied). Satisfaction will be evaluated at the beginning of follow-up visits and after the 6-minute walk test in the ancillary study.
  The question asked will be: "How satisfied are you with the use of the bronchial drainage device to improve your breathlessness?"
Health status | Day 8 (after seven days of intervention).
  Health status will be assessed using the COPD Assessment Test. The CAT score ranges from 0 to 40, with higher values indicating greater impairment of health status. The established minimal clinically important difference for this questionnaire is -2.5 points.
Health related quality of life | Day 8 (after seven days of intervention).
  Quality of life will be assessed using the Saint George's Respiratory Questionnaire. This self-administered questionnaire ranges from 0 to 100, with higher values indicating greater impairment in health-related quality of life. The established minimal clinically important difference for this questionnaire has been established at -4 points.
Use of the intermittent intrapulmonary deflation device | Day 8 (after seven days of intervention).
  Device use will be evaluated through a data collection form that patients will be required to complete after each session. Patients will report the number of sessions per day and the duration of each session.
  Additionally, the number of device uses will be estimated based on consumables, which ensure usage tracking for hygiene reasons and indicate when replacement is necessary.
Adverse events | Day 8 (after seven days of intervention).
  Adverse events occurring during the study, whether related or unrelated to the investigated intervention, will be systematically collected and documented.
Weight of secretions | During visit 1 (day 1).
  Ancillary study. This outcome measure is specific to the ancillary study. The weight of spontaneously expectorated bronchial secretions after the use of the intermittent intrapulmonary deflation device will be assessed over a 1-hour period following the session.
  Saliva will be extracted using a 1 mL micropipette (Pos-D, Mettler Toledo, Viroflay, France), and weight (precision balance, accurate to 0.01 g) of the collected sample will be measured.
Volume of secretions | During visit 1 (day 1).
  Ancillary study. This outcome measure is specific to the ancillary study. The weight of spontaneously expectorated bronchial secretions after the use of the intermittent intrapulmonary deflation device will be assessed over a 1-hour period following the session.
  Saliva will be extracted using a 1 mL micropipette (Pos-D, Mettler Toledo, Viroflay, France), and volume (rounded to the nearest mL using a 1 mL micropipette) of the collected sample will be measured.
Sensory dimension of dyspnea | During visit 1 (day 1).
  Ancillary study. The sensory dimension of dyspnea will be assessed using French version of the Multidimensional Dyspnea Profile questionnaire, taking into account the last 30 seconds of effort during the 6-minute walk test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a greater sensory dimension of dyspnea. The established minimal clinically important difference for this outcome is 2 points.
Affective dimension of dyspnea | During visit 1 (day 1).
  Ancillary study. The affective dimension of dyspnea will be assessed using the french version of the Multidimensional Dyspnea Profile questionnaire, considering the last 30 seconds of effort during the 6-minute walk test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a significant affective dimension of dyspnea. The established minimal clinically important difference for this outcome is 3 points.
Functional exercise capacity - Six-minute walk test | During visit 1 (day 1).
  Ancillary study. Functional exercise capacity will be evaluated using the 6-minute walk test. It will be conducted following the guidelines of the American Thoracic Society and the European Respiratory Society. Patients will be instructed to cover the maximum distance possible within 6 minutes. The test will be performed in a corridor with a minimum length of 30 meters. The established minimal clinically important difference for this test is 25 meters.
Intensity of dyspnea | During visit 1 (day 1).
  Ancillary study. The intensity of dyspnea will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of your breathlessness?" The minimal clinically important difference for this outcome is 1 point. Outcome will be assessed at the end of the six-minute walk test.
Intensity of lower limb fatigue | During visit 1 (day 1).
  Ancillary study. The intensity of muscle fatigue in the lower limbs will be assessed using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of fatigue) and 10 (maximal fatigue). Patients will be asked, "What is the intensity of the fatigue in your legs?" The minimal clinically important difference for this outcome is 1 point. Outcome will be assessed at the end of the six-minute walk test.
Respiratory function - Forced expiratory volume in 1 second | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Vital capacity | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Forced vital capacity | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Ratio between forced expiratory volume in 1 second to forced vital capacity | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France).
Respiratory function - Functional residual capacity | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Total lung capacity | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Residual volume | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France). The values will be expressed liters as well as a percentage of the theoretical values determined by the Global Lung Function Initiative of the European Respiratory Society
Respiratory function - Airway resistance | During visit 1 (day 1).
  Ancillary study. Respiratory function will be evaluated through pulmonary function testing conducted in accordance with international guidelines using a validated plethysmograph (Minibox+TM, PulmOne, Nîmes, France).
Breathing pattern - Tidal volume | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Respiratory rate | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Inspiratory time | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Expiratory time | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Ratio between inspiratory time to expiratory time | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds.
Breathing pattern - Minute ventilation | During visit 1 (day 1).
  Ancillary study. Breathing pattern will be recorded using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) at rest and at the end of the exercise while seated. Data will be acquired via an analog-to-digital converter (Powerlab, AD Instruments, Chalgrove, UK), and the acquisition system will be calibrated before each participant.
  To perform the resting measurements, participants will be fitted with a nose clip and instructed to breathe quietly for a period of five minutes through the pneumotachograph. The most stable minute will be selected for analysis. The measurement will be repeated immediately following the 6-minute walk test over a duration of 30 seconds. Minute ventilation will be calculated as the product of tidal volume and respiratory rate.
Operational lung volume - Inspiratory capacity | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Operational lung volume - End inspiratory lung volume | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  End inspiratory lung volume will be calculated as total lung capacity - inspiratory capacity + tidal volume.
Operational lung volume - End expiratory lung volume | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  End expiratory lung volume will be calculated as total lung capacity - inspiratory capacity.
Critical inspiratory constraints - Ratio between tidal volume to inspiratory capacity | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Critical inspiratory constraints - Ratio between tidal volume to vital capacity | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Critical inspiratory constraints - Inspiratory reserve volume | During visit 1 (day 1).
  Ancillary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
  Inspiratory reserve volume will be calculated as inspiratory capacity - tidal volume.
Critical inspiratory constraints - Ratio between inspiratory reserve volume to total lung capacity | During visit 1 (day 1).
  Ancilary study. Assuming that total lung capacity remains unchanged during exercise, inspiratory capacity will be utilized as a marker of dynamic hyperinflation to estimate operational lung volumes. The measurement of inspiratory capacity will be conducted using a pneumotachograph (MLT1000L, AD Instruments, Oxford, UK) following the same protocols as the assessment of the breathing pattern.
  This measurement will be performed at rest, immediately following the five minutes of calm breathing. Five maximal inspiratory maneuvers will be conducted from functional residual capacity, and the highest value will be used for analysis. The inspiratory capacity measurement will also be repeated immediately after the completion of the 6-minute walk test, with three measurements taken.
Transcutaneous oxygen saturation during a six-minute walk test | During visit 1 (day 1).
  Ancillary study. Transcutaneous oxygen saturation (SpO₂) will be measured at rest and continuously throughout the 6-minute walk test using a pulse oximeter (Nonin WristOx2 3150, Nonin Medical Inc., Plymouth, MN, USA). Data collection will be performed using Nvision software (Henrotch, Aartselaar, Belgium). The SpO₂ value at the end of the test, as well as the nadir SpO₂ (lowest recorded value) during the 6MWT, will be reported. The proportion of patients experiencing oxygen desaturation ≥ 4%, as well as the proportion of patients with desaturation ≥ 4% and SpO₂ < 90%, will also be documented. Finally, the total time spent with SpO₂ < 90% will be analyzed.
Heart rate during the six-minute walk test | During visit 1 (day 1).
  Ancillary study. Heart rate will be measured at rest and continuously throughout the six minute xalk test using a pulse oximeter (Nonin WristOx2 3150, Nonin Medical Inc., Plymouth, MN, USA). Data collection will be performed using Nvision software (Henrotch, Aartselaar, Belgium). The highest HR recorded during the test and the HR at the end of the test will be reported.
Patient satisfaction | During visit 1 (day 1).
  Ancillary study. Patient satisfaction will be assessed using a visual analog scale ranging from 0 (not satisfied at all) to 10 (extremely satisfied). Satisfaction will be evaluated at the beginning of follow-up visits and after the 6-minute walk test in the ancillary study.
  The question asked will be: "How satisfied are you with the use of the bronchial drainage device to improve your breathlessness?"

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Bonnevie, PhD, Principal Investigator — Association ADIR; Francis-Edouard Gravier, PhD, Study Chair — ADIR Association; Antoine Cuvelier, Professor, Study Chair — ADIR Association; Jean-François Muir, Professor, Study Chair — ADIR Association; Astrid Vanheule, Msc student, Study Chair — ADIR Association
Locations (1):
- ADIR Association, Rouen, Normandy, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request for research purposes after publication. This includes de-identified data related to demographic characteristics, as well as endpoints published either in the main manuscript or any supplemental data. Requests should be sent to Dr T. Bonnevie (t.bonnevie@adir-hautenormandie.com).
Supporting Information: SAP
Time Frame: Statistical analysis plan will be made available prior to the commencement of any statistical analysis.
  Individual participant data will be made available after publication.
Access Criteria: Data will be made available upon request, for research purpose. Request should be send to Dr T. Bonnevie (t.bonnevie@adir-hautenormandie.com).

REFERENCES:
- [Background] Ekstrom MP, Bornefalk H, Skold CM, Janson C, Blomberg A, Bornefalk-Hermansson A, Igelstrom H, Sandberg J, Sundh J. Minimal Clinically Important Differences and Feasibility of Dyspnea-12 and the Multidimensional Dyspnea Profile in Cardiorespiratory Disease. J Pain Symptom Manage. 2020 Nov;60(5):968-975.e1. doi: 10.1016/j.jpainsymman.2020.05.028. Epub 2020 Jun 6. PMID 32512047